CLINICAL TRIAL: NCT02136225
Title: Reducing Youth Access to Firearms Through the Health Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-2829; 2013-MU-CX-0002 (Other Grant/Funding Number: National Institute of Justice)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Youth Access to Guns in the Home
Keywords: youth; gun; access; home

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Counseling (Experimental): Intervention: Means restriction counseling. Health care providers will counsel parents on the risks of having a gun, particularly an unlocked gun in the home where youth are present.
  Interventions: Behavioral: Means restriction counseling
- Counseling and locking devices (Experimental): Intervention: Means restriction counseling and locking devices. Health care providers will counsel parents on the risks of having a gun, particularly an unlocked gun, in the home where youth are present. Parents will also receive locking devices to store their guns securely.
  Interventions: Behavioral: Means restriction counseling
- Control group (No Intervention): Youth in the control group will receive usual care.

INTERVENTIONS:
Behavioral: Means restriction counseling — Health care providers will counsel parents on the risks of having a gun, particularly an unlocked gun, in the home where youth are present.
  Arms: Counseling; Counseling and locking devices

SUMMARY:
The purpose of this project is to examine the implementation and effectiveness of an intervention, delivered in a health care setting, to decrease home firearm access by youth. The investigators hypothesize that:

1. parents who receive means restriction education provided by their primary care provider will be more likely to report, at the one month and one year follow-up, that they are storing their guns locked compared to parents who do not receive means restriction counseling.
2. parents who receive a free gun locking device(s) will be more likely to report, at the one month and one year follow-up, that they are storing their guns locked compared to parents who receive means restriction counseling alone;
3. parents whose adolescents are assessed at high risk for violence (> 5 on the Violence Injury Protection and Risk Screen (VIPRS)) or depression (>9 on the Patient Health Questionnaire-9 (PHQ-9)) will be more likely to report storing their gun(s) locked at the one month follow-up compared to parents whose children are assessed as low risk, regardless of whether they receive the counseling alone or counseling plus free locking devices and 4) youth whose parents receive a free gun locking device(s) will be more likely to report less access to guns, at one year follow-up, compared to parents who receive means restriction counseling alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Children's Hospital Colorado in the Adolescent Medicine Clinic
* Scheduled for any type of appointment
* Reports having a gun in the home

Exclusion Criteria:

* Adolescent or parent speaks/reads a language other than English or Spanish
* Adolescent has cognitive disabilities
* Adolescent resides in a group home or detention center

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to one month and one year in the reported number of guns locked in the home. | Baseline, one month, 1 year
  The study examines whether the youth and parents in the treatment groups leads to an increase in the number of guns stored securely (locked) in their home.
Change from baseline to one month and one year in the reported number of locking devices parents use to store their guns. | Baseline, one month, one year
  This study examines whether the youth and parents in the second treatment group, receiving means restriction counseling and locking devices, will increase their use of locking devices compared to youth and parents in the means restriction alone and control groups.

SECONDARY OUTCOMES:
Change from baseline to one month and one year in the number of gun(s) reported locked in their home among parents whose youth are at high risk for violence or depression. | Baseline, one month, one year
  This study examines whether parents whose adolescents are assessed at high risk for violence or depression will be more likely to report, at one month and one year that they are storing their guns locked compared to parents who receive means restriction counseling alone.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sigel, MD, Principal Investigator — University of Colorado, Denver